CLINICAL TRIAL: NCT01327573
Title: Eculizumab Therapy for Chronic Complement-Mediated Injury in Kidney Transplantation: A Randomized, Open-Label, Pilot Intervention Trial
Brief Title: Eculizumab Therapy for Chronic Complement-Mediated Injury in Kidney Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanjay Kulkarni (Other)
Collaborators: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Sanjay Kulkarni, Associate Professor, Yale University
Organization: Yale University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100700716
Record Dates: First submitted 2011-03-30; First posted 2011-04-01 (Estimated); Results first posted 2019-08-12 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-07

CONDITIONS: Kidney; Complications, Allograft
Keywords: chronic kidney allograft injury; complement protein; eculizumab; Kidney transplantation
MeSH Terms: interventions — eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eculizumab (Experimental): eculizumab will be given in addition to standard immunosuppression regimen (oral tacrolimus or equivalent, MMF [mycophenolate mofetil
  ], prednisone)
  Interventions: Drug: eculizumab
- no additional therapy (No Intervention): patients in this arm will receive standard immunosuppression regimen (oral tacrolimus or equivalent, MMF, prednisone only, no additional therapy

INTERVENTIONS:
Drug: eculizumab — * Eculizumab Induction 600mg IV every 7 days for 4 doses
  * Eculizumab 900mg IV 7 days later
  * Eculizumab Maintenance 900mg IV every 14 days for total of 26 weeks
  Other Names: h5G1.1-mAb; Soliris
  Arms: Eculizumab

SUMMARY:
This study is designed to assess the effectiveness of eculizumab in recipients of kidney transplantation with donor-specific antibodies (DSA) and worsening kidney function and to assess if eculizumab improves endothelial cell injury in the kidney.

The investigators hypothesize that complement inhibition with eculizumab will reduce allograft injury, resulting from less complement-mediated injury of endothelial cells and less endothelial cell activation.

DETAILED DESCRIPTION:
This study will address the clinical challenge that currently exists in the management of kidney transplant recipients who have developed de novo DSA, have deteriorating graft function, yet have no established treatment alternative.

This is a randomized, open-label, pilot intervention trial. Post transplant patients with deteriorating renal function (defined as 20% reduction in GFR) will be screened for the development of DSA and biopsied for the presence of C4d deposition. All patients with DSA and those meeting inclusion/exclusion criteria will undergo protocol renal biopsy and will be assessed for C4d deposition. Participants will be randomized to treatment with eculizumab plus standard of care (SOC) or SOC only. Randomization will be stratified by C4d status (C4d+/C4d-) with 10 subjects (7 eculizumab, 3 SOC only) in each stratum.

Eculizumab is an antibody that has been developed to inhibit the complement protein C5. Eculizumab will be delivered via IV according to the following schedule:

* Eculizumab Induction 600mg IV every 7 days for 4 doses
* Eculizumab 900mg IV 7 days later
* Eculizumab Maintenance 900mg IV every 14 days for total of 26 weeks

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recipients greater than 6 months from the date of transplant
* Must be on standard immunosuppression: tacrolimus, mycophenolate mofetil, prednisone and have stable tacrolimus trough levels over past 3 months
* Deteriorating renal function, as defined by 20% reduction in GFR (MDRD calculation)
* Presence of DSA, as defined as MFI > 1100
* Renal biopsy demonstrating no diffuse, irreversible end-stage organ injury (i.e. stage IV Fibrosis)
* Renal biopsy demonstrating C4d deposition (stratum 1) or no C4d deposition (stratum 2)

Exclusion Criteria:

* History of CMV, BK, HSV or other viral infections
* History of chronic, recurrent bacterial infections
* Evidence of tubulitis on renal biopsy or other morphological features of acute cellular rejection or acute humoral rejection
* Renal biopsy demonstrating diffuse, irreversible end-stage organ injury
* Absolute GFR < 25 (MDRD calculation)
* Inability to provide informed consent
* History of poor vascular access
* Refusal to use double barrier contraception during study participation
* Patients actively enrolled in other clinical trials

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Kulkarni, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

REFERENCES:
- [Background] Terasaki PI, Ozawa M. Predicting kidney graft failure by HLA antibodies: a prospective trial. Am J Transplant. 2004 Mar;4(3):438-43. doi: 10.1111/j.1600-6143.2004.00360.x. PMID 14961999
- [Background] Worthington JE, McEwen A, McWilliam LJ, Picton ML, Martin S. Association between C4d staining in renal transplant biopsies, production of donor-specific HLA antibodies, and graft outcome. Transplantation. 2007 Feb 27;83(4):398-403. doi: 10.1097/01.tp.0000251430.11723.b6. PMID 17318071
- [Background] Al-Lamki RS, Bradley JR, Pober JS. Endothelial cells in allograft rejection. Transplantation. 2008 Nov 27;86(10):1340-8. doi: 10.1097/TP.0b013e3181891d8b. PMID 19034000
- [Background] Brodsky RA, Young NS, Antonioli E, Risitano AM, Schrezenmeier H, Schubert J, Gaya A, Coyle L, de Castro C, Fu CL, Maciejewski JP, Bessler M, Kroon HA, Rother RP, Hillmen P. Multicenter phase 3 study of the complement inhibitor eculizumab for the treatment of patients with paroxysmal nocturnal hemoglobinuria. Blood. 2008 Feb 15;111(4):1840-7. doi: 10.1182/blood-2007-06-094136. Epub 2007 Nov 30. PMID 18055865
- [Background] Davin JC, Gracchi V, Bouts A, Groothoff J, Strain L, Goodship T. Maintenance of kidney function following treatment with eculizumab and discontinuation of plasma exchange after a third kidney transplant for atypical hemolytic uremic syndrome associated with a CFH mutation. Am J Kidney Dis. 2010 Apr;55(4):708-11. doi: 10.1053/j.ajkd.2009.08.011. Epub 2009 Oct 25. PMID 19854549

RESULTS

PARTICIPANT FLOW:
Groups:
- Eculizumab: eculizumab will be given in addition to standard immunosuppression regimen (oral tacrolimus or equivalent, MMF [mycophenolate mofetil
  ], prednisone)
  eculizumab: • Eculizumab Induction 600mg IV every 7 days for 4 doses
  * Eculizumab 900mg IV 7 days later
  * Eculizumab Maintenance 900mg IV every 14 days for total of 26 weeks
Period: Overall Study
Arm/Group | Eculizumab | no Additional Therapy
Started | 11 | 5
Received Treatment/Control as Allocated | 10 | 5
Completed | 8 | 4
Not Completed | 3 | 1
Not completed — Physician Decision | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eculizumab | no Additional Therapy | Total
Number analyzed (Participants) | 10 | 5 | 15
Age, Continuous [Median (Full Range); unit: years] | 38 [20 to 57] | 44 [33 to 65] | 43 [20 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 7 | 2 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 6 | 2 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 10 | 5 | 15
C4d Status at Randomization [Number; unit: participants]
  Positive | 5 | 1 | 6
  Negative | 5 | 4 | 9
Baseline DSA (Donor Specific Antibody) MFI (mean fluorescent intensity) [Median (Full Range); unit: MFI] — The mean fluorescent intensity of the DSA (donor specific antibody) is derived per participant.
  Median and full range values for each arm are reported here.
  MFI | 5,000 [2,900 to 13,400] | 3,100 [1,100 to 6,000] | 4,600 [1,100 to 13,400]

OUTCOME MEASURES:

1. Primary Outcome: Baseline eGFR (Estimated Glomerular Filtration Rate)
Time Frame: Baseline
Measure: Mean (95% Confidence Interval); unit: mL/min/1.73 m2
Arm/Group | Eculizumab | no Additional Therapy
Number analyzed (Participants) | 10 | 5
mL/min/1.73 m2 | 30.04 [23.77 to 36.31] | 30.04 [23.77 to 36.31]

2. Primary Outcome: Estimated Glomerular Filtration Rate (eGFR) at Months 2,3,4,5,6
Description: Primary statistical analysis of change from baseline was conducted with mixed effects modeling providing calculated estimates.
Time Frame: Months 2,3,4,5,6
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/min/1.73 m2
Arm/Group | Eculizumab | no Additional Therapy
Number analyzed (Participants) | 10 | 5
mL/min/1.73 m2
  Month 2 | 29.34 [26.61 to 32.07] | 31.34 [27.45 to 35.24]
  Month 3 | 29.56 [26.56 to 32.55] | 30.68 [26.43 to 34.93]
  Month 4 | 29.78 [26.43 to 33.13] | 30.02 [25.29 to 34.75]
  Month 5 | 29.99 [26.23 to 33.76] | 29.35 [24.06 to 34.65]
  Month 6 | 30.21 [25.98 to 34.44] | 28.69 [22.77 to 34.61]
Statistical Analysis 1: Comparison: Eculizumab vs no Additional Therapy; Analysis used eGFR, group, time, and group-by-time variables; Test type: Superiority or Other; p = 0.09, Mixed effects model analysis — This p-value was for the overall slope difference between groups (i.e. the interaction between group and time). Significance level was set at 0.1 a priori

3. Primary Outcome: Group Difference Percentage Change in 6-month Estimated Glomerular Filtration Rate (eGFR)
Description: These data were calculated by mean 6-month eGFR minus baseline mean eGFR divided by baseline eGFR. Presented below are the between groups results. These results were derived from the results in the outcome "Estimated Glomerular Filtration Rate (eGFR) at Months 2,3,4,5,6".
Time Frame: 6 months
Population: These are the between groups percent change that represents the difference between groups when controlling for baseline. Outcome measure #2 provides the data by treatment arm where these data are derived.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage change
Groups:
- Between Groups Difference: These are the percent change between group differences derived from the Estimated Glomerular Filtration Rate (eGFR) at Months 2,3,4,5,6 outcome.
Arm/Group | Between Groups Difference
Number analyzed (Participants) | 16
percentage change
  Month 2 | 6.66 [-9.21 to 22.53]
  Month 3 | 3.73 [-13.62 to 21.08]
  Month 4 | 0.80 [-18.52 to 20.12]
  Month 5 | -2.13 [-23.77 to 19.51]
  Month 6 | -5.06 [-29.28 to 19.16]

ADVERSE EVENTS:
Arm/Group | Eculizumab | no Additional Therapy
Serious Adverse Events (participants affected / at risk) | 4/10 | 3/5
Other Adverse Events (participants affected / at risk) | 2/10 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eculizumab (N=10) | no Additional Therapy (N=5)
Graft Failure (Renal and urinary disorders) | 2 (2) | 1 (1)
Bacterial Infection (Infections and infestations) | 1 (1) | 1 (1)
Viral Infection (Infections and infestations) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eculizumab (N=10) | no Additional Therapy (N=5)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Viral Infection (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less